CLINICAL TRIAL: NCT02109731
Title: Upper Airway Physical Therapy for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Suzanne Karan, Principal investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24149
Record Dates: First submitted 2012-02-09; First posted 2014-04-10 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome (OSAS); Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Negative airway pressure delivery (Experimental): Negative airway pressure delivery (breathing against a vaccuum) in order to improve the tone of the upper airway muscles and make them less susceptible to collapse during sleep.
  Interventions: Other: Negative airway pressure delivery

INTERVENTIONS:
Other: Negative airway pressure delivery — Negative airway pressure delivery (breathing against a vaccuum) in order to improve the tone of the upper airway muscles and make them less susceptible to collapse during sleep.

SUMMARY:
The purpose of this study is to determine the effectiveness and feasibility of upper airway muscle physical therapy utilizing negative airway pressure (NAP) breathing training in patients with Obstructive Sleep Apnea Syndrome (OSAS) in reducing both signs (apnea hypopnea index) and symptoms (i.e., daytime sleepiness).The key to the proposed therapy is the use of Negative Air Pressure when awake so that the increased reflex phasic drive to the muscles will result in muscle conditioning. Interestingly, other studies have indicated that upper airway muscle training may be useful in treating OSAS, but these studies used techniques that were not scientifically designed{Puhan, 2006 8195 /id} or used a technique (electrical stimulation) that was not well tolerated.{Lequeux, 2005 7514 /id}

DETAILED DESCRIPTION:
Overview: Subjects with OSAS (but not using continuous positive airway pressure CPAP) will undergo NAP physical therapy of the upper airway, utilizing a physiologically determined training pressure and protocol, three days a week (approximately 30 minute sessions each) for a period of three months. Overnight sleep studies (PSGs) will be performed pre- and post-study. Primary outcome measurements include the pre- and post-study Apnea/Hypopnea index (AHI) and daytime hypersomnolence symptom scores. Each subject's total study time is approximately a 3-4 month period which includes screening visit, pre and post study overnight polysomnography, and therapy sessions of 3-4 a week for three months.

ELIGIBILITY:
Inclusion Criteria:

18 and over and any persons who have been diagnosed with OSAS (AHI over 15) and who are not utilizing CPAP

Exclusion Criteria:

Participants will be excluded if: Pregnant, Breastfeeding or any bleeding abnormalities, there is a major upper airway morphologic abnormality (e.g., retrognathia, Pierre-Robin syndrome), they have had any airway surgery (except tonsillectomy as a child),they regularly use any drugs that are known to depress the central nervous system (such as benzodiazepines, narcotics), they consume 14 alcoholic drinks a week or 2 a day,they are undergoing a current or planned intervention for weight reduction or are morbidly obese (body mass index 40 kg/m2), or they have any unstable medical or psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Karan, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative Airway Pressure Delivery
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects have a diagnosis of OSA and are not currently receiving CPAP therapy
Arm/Group | Negative Airway Pressure Delivery
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
BMI [Mean (Standard Deviation); unit: kilograms per meter squared] | 32.9 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Delta of Apnea Hypopnea Index (AHI) as Measured by Polysomnography (PSG)
Description: The pre-study AHI (before the NAP treatment was applied) was measured and quantified and compared to the post study AHI (after three months of NAP treatment) and the difference between pre and post therapy is reported. The AHI is an hourly rate of breathing disturbance (apneas and hypopneas per hour) that is calculated while subjects are evaluated during an overnight sleep study, with polysomnography applied (PSG). For example, while a subject is spending the night in the PSG laboratory sleeping, his/her breathing is evaluated for evidence of apneas and hypopneas during various stages of sleep. Sleep is measured with electroencephalography. And breathing is measure with respiratory excursions via chest/abdominal plethysmography recordings and airflow from the nose/mouth.
Time Frame: three months
Population: subjects with a diagnosis of OSA
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Negative Airway Pressure Delivery
Number analyzed (Participants) | 15
events per hour | 4.27 (11.96)

ADVERSE EVENTS:
Arm/Group | Negative Airway Pressure Delivery
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No